CLINICAL TRIAL: NCT03115970
Title: Feasibility of Lactate Level Evaluation in Prehospital Care in Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Marcela Bilska, Dr., Masaryk Hospital Usti nad Labem
Other Study IDs: KAPIM-L
Record Dates: First submitted 2017-04-09; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Trauma, Multiple; Lactate Blood Increase
MeSH Terms: conditions — Multiple Trauma; Hyperlactatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients: All patients having / suspected to have severe trauma injuries
  Interventions: Procedure: capillary and venous lactate level measurement

INTERVENTIONS:
Procedure: capillary and venous lactate level measurement — capillary and venous lactate level measurement

SUMMARY:
Capillary or venous lactate level evaluation in prehospital care could be simple and beneficial tool for optimising prehospital care in patients with severe trauma.

DETAILED DESCRIPTION:
Evaluation of blood lactate level and its trend are important morbidity and mortality predictive factors. In prehospital care, lactate level is more sensitive marker and have better prognostic value in severe trauma than basic vital signs. Worse outcome is associated with levels between 2 - 4 mmol/l. Measurement of lactate level in venous or capillary blood is quick and simple method with minimal risks and with no special needs for medical staff training. In spite of good availability of this method in the Czech Republic the method feasibility has never been analysed in patients with severe trauma.

ELIGIBILITY:
Inclusion Criteria:

* patient having / suspected to have severe trauma treated by cooperating Emergency Medical System organization

Exclusion Criteria:

* possible alterations of plasma lactate level in the time of trauma (seizure, malignity, use of beta-2 agonists, severe liver and/or kidney failure, ketoacidosis, intoxication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having / suspected to have severe trauma
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of lactate level measurement | 1 day - the time the patient is treated by Emergency Medical System
  Proportion of subjects with measured and recorded prehospital lactate level

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Bilska, Dr., Principal Investigator — Masaryk Hospital in Usti nad Labem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kruse O, Grunnet N, Barfod C. Blood lactate as a predictor for in-hospital mortality in patients admitted acutely to hospital: a systematic review. Scand J Trauma Resusc Emerg Med. 2011 Dec 28;19:74. doi: 10.1186/1757-7241-19-74. PMID 22202128
- [Background] Jansen TC, van Bommel J, Mulder PG, Rommes JH, Schieveld SJ, Bakker J. The prognostic value of blood lactate levels relative to that of vital signs in the pre-hospital setting: a pilot study. Crit Care. 2008;12(6):R160. doi: 10.1186/cc7159. Epub 2008 Dec 17. PMID 19091118
- [Background] Pearse RM. Extending the role of lactate measurement into the prehospital environment. Crit Care. 2009;13(1):115. doi: 10.1186/cc7687. Epub 2009 Feb 10. PMID 19232076
- [Background] Rossaint R, Bouillon B, Cerny V, Coats TJ, Duranteau J, Fernandez-Mondejar E, Filipescu D, Hunt BJ, Komadina R, Nardi G, Neugebauer EA, Ozier Y, Riddez L, Schultz A, Vincent JL, Spahn DR. The European guideline on management of major bleeding and coagulopathy following trauma: fourth edition. Crit Care. 2016 Apr 12;20:100. doi: 10.1186/s13054-016-1265-x. PMID 27072503